CLINICAL TRIAL: NCT04199793
Title: Assessment of Lavare Cycle Implementation Among Patients Following HeartWare Left Ventricular Assist Device Implantation: A Prospective Randomized Controlled Pilot Study
Brief Title: Lavare Cycle in Patients Receiving HeartWare Left Ventricular Assist Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The device (HeartWare) was recalled and discontinued by the FDA
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sandip Zalawadiya, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HeartWareLavare1
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Results first posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-11

CONDITIONS: Thromboembolism; Hemolysis; Stroke
Keywords: Lavare Cycle; HeartWare LVAD; Thromboembolic events
MeSH Terms: conditions — Thromboembolism; Hemolysis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Lavare Cycle On (Active Comparator): For the patients randomized to "Lavare On" group, the Lavare™ cycle will be turned on upon device interrogation after patients return to intensive care unit from the operating room.
  Interventions: Device: Lavare On
- Lavare Cycle Off (Active Comparator): For the patients randomized to "Lavare Off" group, the Lavare™ cycle will be turned off upon device interrogation after patients return to intensive care unit from the operating room.
  Interventions: Device: Lavare Off

INTERVENTIONS:
Device: Lavare On — For the patients randomized to "Lavare On" group, the Lavare™ cycle will be turned on upon device interrogation after patients return to intensive care unit from the operating room.
  Arms: Lavare Cycle On
Device: Lavare Off — For the patients randomized to "Lavare Off" group, the Lavare™ cycle will be turned off upon device interrogation after patients return to intensive care unit from the operating room.
  Arms: Lavare Cycle Off

SUMMARY:
Left ventricular assist device (LVAD) patients remain at risk for pump thrombus and thromboembolic events through multiple mechanisms. The HeartWare® Ventricular Assist System (HVAD®, HeartWare Inc., Framingham, MA, USA) includes a novel speed modulation feature called Lavare™ cycle. The Lavare™ Cycle is aimed to promote washing of left ventricle to decrease blood stasis and subsequent risk of thrombus formation, ingestion and/or expulsion. No prior study has prospectively evaluated the impact of Lavare™ cycle on patient outcomes in a randomized fashion. We intend to assess effects of Lavare™ Cycle among patients receiving HVAD LVAD in this randomized controlled pilot project.

DETAILED DESCRIPTION:
Left ventricular assist device (LVAD) patients remain at risk for pump thrombus and thromboembolic events through multiple mechanisms. The HeartWare® Ventricular Assist System (HVAD®, HeartWare Inc., Framingham, MA, USA) includes a novel speed modulation feature called Lavare™ cycle. It consists of 3 phases: phase 1 - a 200 rpm decrease from baseline speed for 2 seconds, phase 2 - a 100 rpm increase from baseline for 1 second and phase 3 - return of speed to baseline; this cycle repeats itself once every minute.

The LavareTM Cycle is aimed to promote washing of left ventricle to decrease blood stasis and subsequent risk of thrombus formation, ingestion and/or expulsion. In a post-hoc analysis of ReVOLVE registry, which includes 248 patients implanted with the HVAD following Conformité Européenne Mark in nine centers in Europe and Australia, no adverse impact on survival was observed with Lavare™ cycle. Additionally, lower risk of stroke, sepsis and right heart failure was observed among those with Lavare™ cycle in the above-mentioned study. However, no prior study has prospectively evaluated the impact of Lavare™ cycle on patient outcomes in a randomized fashion. In this prospective randomized controlled trial, we intend to assess the role of Lavare™ cycle in pump related complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Approved for or supported with HeartWare durable LVAD
3. Capable of giving informed consent

Exclusion Criteria:

1. For those undergoing new device implantation:

   1. Age <18 years
   2. Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) profile 1 at the time of implantation
   3. Presence of intra-cardiac thrombus
   4. History of thromboembolic event within previous 3 months of enrollment
2. For those with prior LVAD implantation with on-going support:

   1. Support duration <3 months
   2. History of prior LVAD pump exchange
   3. History of LVAD pump hemolysis or thrombosis as defined by INTERMACS criteria
   4. History of stroke or transient ischemic event within previous 3 months of enrollment
   5. History of post-LVAD severe right ventricular failure as defined by INTERMACS criteria within previous 3 months of enrollment
   6. History of pump-related infection treated within previous 3 months of enrollment or those on chronic antibiotics suppressive therapy for pump related infection
   7. History of post-LVAD intra-cardiac or arterial thrombus or thromboembolic event within previous 3 months of enrollment
   8. International Normalized Ratio (INR) <2 within previous 30-days from the date of enrollment
   9. Aspirin dose <325 mg/day
   10. Lactate Dehydrogenase (LDH) levels ≥ 3 times the upper normal limit in previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Zalawadiya, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St Vincent Hospital Indianapolis, Indianapolis, Indiana
  - Vanderblt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zimpfer D, Strueber M, Aigner P, Schmitto JD, Fiane AE, Larbalestier R, Tsui S, Jansz P, Simon A, Schueler S, Moscato F, Schima H. Evaluation of the HeartWare ventricular assist device Lavare cycle in a particle image velocimetry model and in clinical practice. Eur J Cardiothorac Surg. 2016 Nov;50(5):839-848. doi: 10.1093/ejcts/ezw232. Epub 2016 Sep 7. PMID 27605222

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants signed informed consent. One patient was not randomized due to improved health. Total of 8 patients were randomized.
Period: Overall Study
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Started | 4 | 4
Completed | 1 | 1
Not Completed | 3 | 3
Not completed — Sponsor Withdrew the device off market; study stopped | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lavare Cycle On | Lavare Cycle Off | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [50 to 62] | 54.5 [52.5 to 57] | 54.5 [51.7 to 58.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint of Total Ischemic Events, Thromboembolic Events, Pump Hemolysis or Thrombosis, Pump Exchange
Description: INTERMACS definitions of cerebrovascular events, pump hemolysis/ thrombosis will be used. Pump malfunction needing device exchange or emergent transplant will also be included in the main composite event
Time Frame: 6 months
Population: Data analysis was not completed because only one participant completed each arm and showing data could violate privacy interests. The department also did not allocate resources for further analysis as the trial was terminated early and was missing sufficient samples and data points for the prespecified analysis.
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: All-cause Mortality
Description: death from any cause
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Survival to Transplantation
Description: Number of days supported on LVAD until transplant
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Rehospitalizations
Description: Any cardiac and non-cardiac re-hospitalizations since trial enrollment
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mucosal Bleeding
Description: Epistaxis, gastrointestinal bleeding, urological bleeding events will be analyzed
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Right Ventricular Failure
Description: INTERMACS definitions for Right ventricular failure will be analyzed
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Device Related Infection
Description: LVAD device systems related infections will be analyzed
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Aortic Insufficiency
Description: Echocardiographic evidence will be used to define severity of aortic insufficiency
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in 6 Minute Walk Test
Description: The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Changes in New York Heart Association Class
Description: Functional class will be assessed at baseline and during follow up to assess improvement in functional status
Time Frame: Baseline to 6 months
Population: as for outcome 1
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Quality of Life Measured by The Kansas City Cardiomyopathy Questionnaire
Description: Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The score can range from 0-100, in which higher scores reflect better health status.
Time Frame: 6 months
Population: as for outcome 1
Arm/Group | Lavare Cycle On | Lavare Cycle Off
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 180-days
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse events were collected from the time of randomization through participant completion.
Arm/Group | Lavare Cycle On | Lavare Cycle Off
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4 | 4/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lavare Cycle On (N=4) | Lavare Cycle Off (N=4)
Rehospitalization due to low INR (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Rehospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pneumothorax requiring chest tube placement; Need for inotropic support during hospitalization.
Rehospitalization (Surgical and medical procedures) | 0 (0) | 1 (1) — Surgical wound dehiscence requiring wound vac placement
Rehospitalization (Infections and infestations) | 0 (0) | 1 (1) — Infections of the genitourinary, gastrointestinal and pulmonary systems.
Right heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Rehospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) — Colitis
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) — Required medications (anti-arrhythmic) adjustments
Pump/Drive line infection (Infections and infestations) | 0 (0) | 2 (2)
Other systems infections (Infections and infestations) | 0 (0) | 2 (2) — Not requiring hospitalizations
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Device malfunction alarms (Surgical and medical procedures) | 1 (1) | 1 (1) — Includes controller exchange

LIMITATIONS AND CAVEATS:
The study was terminated early due to the sponsor withdrew the device off market.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT04199793/Prot_SAP_000.pdf